CLINICAL TRIAL: NCT01291810
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Clinical Efficacy, Safety and Immunogenicity of Neovacs' TNFα-Kinoid in Adult Subjects With Crohn's Disease
Brief Title: Clinical Efficacy of TNFa Kinoid in Crohn's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neovacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNF-K-005
Record Dates: First submitted 2010-12-17; First posted 2011-02-08 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TNF Kinoid (Experimental)
  Interventions: Biological: TNF Kinoid
- Placebo (Placebo Comparator)
  Interventions: Biological: WFI

INTERVENTIONS:
Biological: TNF Kinoid — TNF Kinoid
  Arms: TNF Kinoid
Biological: WFI — WFI
  Arms: Placebo

SUMMARY:
The safety and immunogenicity of the TNFα-Kinoid (TNF-K) have been evaluated in a phase I-II clinical study conducted in subjects with Crohn's Disease (CD). Preliminary results of clinical efficacy are promising.

The principal aim of the present study is to confirm the clinical efficacy of the TNF-K in subjects with moderate to severe CD. Subjects with secondary resistance or intolerance to anti-TNFα monoclonal antibodies will be enrolled in this trial. In addition, the immune responses and the safety elicited by TNF-K will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 65 years, inclusive.
2. Have had a diagnosis of Crohn's disease for at least 6 months.
3. Moderate to severe active Crohn's disease defined as a Crohn's Disease Activity Index (CDAI) score ≥ 220 and ≤ 450, and presence of colonic mucosal ulcerations in at least 2 segments, or ulcerations on ≥ 10% of the mucosal surface if only one segment is involved.
4. Have developed secondary resistance to anti-TNFα therapy.

Exclusion Criteria:

1. Primary non-response to a previously received treatment directed against TNFα Or Intolerance related to the primary pharmacological effect of anti-TNFα such as for instance, but not limited to, severe or opportunistic infections and demyelinating or autoimmune diseases.
2. History of severe systemic bacterial, fungal, viral, or parasitic infections within the 3 months prior to screening; or the occurrence of any acute infection within 2 weeks of the first administration of study drug.
3. Treatment with immunosuppressive or immunomodulatory drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Clinical remission, defined as a CDAI score ≤ 150 points at week 8. | Week 8

SECONDARY OUTCOMES:
Clinical responses, defined as a decrease of at least 70 points (CDAI-70) and at least 100 points (CDAI-100) in the CDAI score at week 8 vs baseline | week 8
Endoscopic response, defined as a reduction of at least 50% in the Crohn's Disease Endoscopic Index of Severity (CDEIS) score or in the Simple Endoscopic Score for Crohn's Disease (SES-CD) at week 12 vs baseline | week 12
Biological response as defined by a decrease or normalization of calprotectin levels in stools | Week 12
Safety assessments will be conducted throughout the study and will include physical examinations, vital signs, 12-lead electrocardiograms (ECGs), clinical laboratory evaluations, and the recording of adverse events (AEs). | Week 28
Immunogenicity: o Anti-TNFα antibodies by Enzyme-Linked Immunosorbent Assay (ELISA) o Anti-TNFα neutralizing antibody activity o Anti-KLH antibodies by ELISA | week 12

CONTACTS AND LOCATIONS:
Locations (58):
- Belgium (4):
  - Imelda Clinic, Bonheiden
  - Cliniques Universitaires St Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Katholiek Unversiteit van Leuven, Leuven
- Bulgaria (7):
  - University Multiprofile Hospital St. Georgi, Plovdiv
  - Alexandrovska University Hospital, Sofia
  - Medical Institute- Ministry of Interior Clinic of Gastroenterology, Sofia
  - MMA Clinic of Gastroenterology, Sofia
  - UMHAT "St. Ivan Rilsky", Sofia
  - UMHAT Queen Yoanna - ISUL, Sofia
  - Clinic of Gastroenterology/ University Hospital Varna, Varna
- Croatia (4):
  - Clinical Hospital Centre Rijeka, Rijeka
  - General Hospital Zadar, Zadar
  - Clinical Hospital Centre Zagreb,, Zagreb
  - University Hospital Dubrava, Zagreb
- Czechia (3):
  - Faculty Hospital in Hradec Králové, Hradec Králové
  - Faculty Hospital Olomouc, Olomouc
  - IBD Clinical and Research Centre, Prague
- France (12):
  - CHU Hôpital Nord, Amiens
  - Hôpital Haut-Lévêque, Bordeaux
  - CHU Caen, Caen
  - CHU Côte de Nacre, Caen
  - Hopital Beaujon (APHP), Clichy
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital A Huriez CHRU Lille, Lille
  - CHU Nancy Hôpital Brabois, Nancy
  - CHU de Nice Hôpital de l'Archet, Nice
  - Hôpital St Louis, Paris
  - CHU Rouen, Rouen
  - CHU Rangueil, Toulouse
- Germany (18):
  - Charité Campus Virchow-Klinikum, Berlin
  - Gastroenterologische Spezialpraxis, Berlin
  - Klinik mit Schwerpunkt Gastroenterologie, Campus Charité Mitte, Berlin
  - Klinikum Braunschweig, Braunschweig
  - Abteilung Innere Medizin Evangelisches Krankenhaus Kalk gGmbH, Cologne
  - Klinik für Allg. Innere Medizin, Gastroenterologie und Diabetologie, Kliniken-Essen-Mitte/Evang. Huyssenstiftung, Essen
  - Universitätsklinik und Poliklinik für Innere Medizin I, Halle
  - Asklepios Westklinikum Hamburg, Hamburg
  - Hamburgisches Forschungsinstitut für CED, Hamburg
  - I. Medizinische Klinik und Poliklinik, Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - Gastroenterologische Gemeinschaftspraxis im Ärztehaus am Ev. Krankenhaus Herne, Herne
  - Klinik für Innere Medizin II Abteilung Gastroenterologie, Hepatologie, Infektiologie, Jena
  - Klinik für Innere Medizin I, Kiel
  - Internistische Gemeinschaftspraxis für Verdauungs- und Stoffwechselkrankheiten, Leipzig
  - I. Med. Klinik und Poliklinik, Mainz
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Ulm, Ulm
- Hungary (3):
  - Fővárosi Önkormányzat Péterfy Sándor utcai Kórháza, Budapest
  - Semmelweis Egyetem ÁOK, Budapest
  - DE OEC, Debrecen
- Netherlands (2):
  - Academic Medical Center (AMC), Amsterdam
  - Free University Medical Centre in Amsterdam (VUMC), Amsterdam
- Romania (5):
  - Colentina Clinical Hospital, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Mediclass Sananova SRL, Bucharest
  - Dr. Citu Outpatient Clinic, Timișoara
  - Polyclinic Private Practice Algomed SRL, Timișoara